CLINICAL TRIAL: NCT03895086
Title: Fibromyalgia and Specific Physical Activity
Acronym: FibrAPSpé
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: impossible enrollement
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHD110-18
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific Physical Activity (Experimental): Specific patient care in telephone coaching of fibromyalgia patients.
  Interventions: Other: Specific Physical Activity
- Classic Physical Activity (Other): Classic patient care in common group of multipathological patients.
  Interventions: Behavioral: Classic Physical Activity

INTERVENTIONS:
Other: Specific Physical Activity — An individual one hour face-to-face session conducted by adaptated physical activities teachers followed by eight telephone sessions by physical therapists and adaptated physical activities teachers (4 sessions each)
  Arms: Specific Physical Activity
Behavioral: Classic Physical Activity — One session per week in groups conducted by adaptated physical activities teachers of "Siel Bleu" association
  Arms: Classic Physical Activity

SUMMARY:
Fibromyalgia is a common, expensive and controversial condition, one of whose origins would be central nervous system sensitization to pain.

Usual treatment consists of multimodal care including physical activity. This dosage should be adapted to the patient's health needs. Currently recommended physical exercise is aerobic work associated with muscle reinforcement, without evidence of superiority of the efficacy of one over the other. Recommended dosage for aerobic exercises is 20 minutes (or twice 10 minutes), two to three times a week (70 - 80% of Theoretical Maximum Heart Rate).

At the Vendee Departmental Hospital Center (CHD), adapted physical activity is proposed to fibromyalgia patientsby the associative group "Siel Bleu". This physical activity, performed with patients suffering from different pathologies, is non specific for fibromyalgia context.

In parallel, a preliminary study showed the interest of a lifestyle coaching for fibromyalgia patients, performed by physiotherapists, nurses and coaches specifically trainede.

Another possibility seems to be personalized coaching with a physical activity adapted to the physical and organizational constraints of the patient, and specific to pathology. This solution would make it possible to adapt to the patient's choice of physical activities, to ensure a better adaptation to their physical and organizational constraints as well as a better individualized follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient whose FIQ ≤ 59/100
* Patient who can be followed for 12 months in the CETD
* Patient able to follow the adaptated physical activities proposed by "Siel Bleu", on the physical and organizational level
* Patient with a smartphone and/or a computer (mac/pc) with an internet connection allowing the use of a tracking application linked to the activity tracker
* Patient with the ability to understand protocol and consenting to participate in this study
* Patient benefiting from a social cover

Exclusion Criteria:

* Patient participating in an interventional trial within 3 months of enrollment
* Pregnant or lactating woman, or having the possibility to procreate without effective contraception
* Patient minor, under guardianship, curators or deprived of liberty
* Patient unable to follow the protocol, according to the judgment of the investigator, or refusing to use of digital applications
* Patient with contraindications to physical activity
* Patient having already followed the physical activities proposed by 'Siel Bleu"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas RULLEAU, Principal Investigator — CHD Vendée
Locations (2):
- France (2):
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier Universitaire, Nantes

REFERENCES:
- [Background] Rulleau T, Planche L, Etcheverrigaray F, Dorion A, Kacki N, Miot M, Liaigre A, Ganem Y, Schmidt A, Taddei F, Acapo S, Nizard J, Pluchon YM. Comparison of patient-led, fibromyalgia-orientated physical activity and a non-specific, standardised 6-month physical activity program on quality of life in individuals with fibromyalgia: a protocol for a randomised controlled trial. Trials. 2020 Sep 17;21(1):800. doi: 10.1186/s13063-020-04730-3. PMID 32943085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 1 participant was randomized to the treatment
Period: Overall Study
Arm/Group | Specific Physical Activity | Classic Physical Activity
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Early termination study | 1 | 0

BASELINE CHARACTERISTICS:
Population: early termination study
Groups:
- Total: Total of all reporting groups
Arm/Group | Specific Physical Activity | Classic Physical Activity | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Data not collected - study stopped prematurely
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 0
  Male |  |  | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Compare the Interest of a Specific Physical Activity Program on Patients' Quality of Life
Description: Evolution of the Fibromyalgia Impact Questionnaire (FIQ) score (questionnaire of specific quality of life in the management of fibromyalgia patients) between the beginning of care (J0) and six months (M6).
  The scale score ranges from 0 to 100. The higher the score, the greater the difficulty in functioning and the severity of symptoms.
Time Frame: 6 months after randomization
Population: Only one patient was enrolled in the study - data was not collected
Arm/Group | Specific Physical Activity | Classic Physical Activity
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Death, serious adverse events and other (non serious adverse events) were not assessed for the study
Arm/Group | Specific Physical Activity | Classic Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT03895086/Prot_SAP_000.pdf